CLINICAL TRIAL: NCT02846883
Title: Mesenchymal Stem Cells Induce Regulatory T Cells in Patients With Aortic Aneurysm
Brief Title: Safety and Efficacy of Allogeneic MSCs in Promoting T-regulatory Cells in Patients With Small Abdominal Aortic Aneurysms
Acronym: VIVAAA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Early Termination as required by VA DSMB due to slow enrollment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLNB-06-15F; 1510579216 (Other: IU IRB); NCT02843854 (obsolete NCT alias)
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: aneurysms; aortic aneurysm; Abdominal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm; Aortic Aneurysm | interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intravenous infusion of 1 million allogenic MSCs/kg (Active Comparator): In a randomized fashion, the MSCs, in the appropriate dose, will be shipped to the performance site where the MSCs will be thawed, diluted and administered. The thawed MSCs with be administered within 4 hours to subjects in a monitored setting with telemetry and pulse oximetry. Patients will be premedicated with hydrocortisone and diphenhydramine. All subjects will be monitored throughout the infusion procedure with vital signs and pulse oximetry at 15 minutes prior to infusion and ending 2 hours post procedure. They will also be evaluated for clinical signs of pulmonary distress. Subjects will be discharged 2 hours post-infusion if no signs of complications.
  Interventions: Biological: 1 million MSCs/kg
- Intravenous infusion of 3 million allogeneic MSCs/kg (Active Comparator): In a randomized fashion, the MSCs, in the appropriate dose, will be shipped to the performance site where the MSCs will be thawed, diluted and administered.The thawed MSCs with be administered within 4 hours to subjects in a monitored setting with telemetry and pulse oximetry. Patients will be premedicated with hydrocortisone and diphenhydramine. All subjects will be monitored throughout the infusion procedure with vital signs and pulse oximetry at 15 minutes prior to infusion and ending 2 hours post procedure. They will also be evaluated for clinical signs of pulmonary distress. Subjects will be discharged 2 hours post-infusion if no signs of complications.
  Interventions: Biological: 3 million MSCs/kg
- Intravenous infusion of Plasmalyte A (placebo) (Placebo Comparator): In a randomized fashion, the Plasmalyte A will be shipped to the performance site where it will be thawed and administered. The Plasmalyte A will be administered within 4 hours to subjects in a monitored setting with telemetry and pulse oximetry as will be performed on active groups in order to protect the blinding of this study. Patients will be pre-medicated with hydrocortisone and diphenhydramine. All subjects will be monitored throughout the infusion procedure with vital signs and pulse oximetry at 15 minutes prior to infusion and ending 2 hours post procedure. They will also be evaluated for clinical signs of pulmonary distress. Subjects will be discharged 2 hours post-infusion if no signs of complications.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: 1 million MSCs/kg — Intravenous infusion of 1 million allogeneic MSCs/kg.
  Arms: Intravenous infusion of 1 million allogenic MSCs/kg
Biological: 3 million MSCs/kg — Intravenous infusion of 3 million allogeneic MSCs/kg
  Arms: Intravenous infusion of 3 million allogeneic MSCs/kg
Drug: Placebo — Intravenous infusion of Plasmalyte A (placebo)
  Other Names: Plasmalyte A
  Arms: Intravenous infusion of Plasmalyte A (placebo)

SUMMARY:
This project is to determine the safety and explore the effectiveness of allogeneic (not cells of the participant but those of another human) mesenchymal stromal cells (MSCs) in decreasing inflammation and possible enlargement of the participants' abdominal aortic aneurysm. Participants will be selected as a possible subject because of an abdominal aortic aneurysm discovered on the ultrasound or computed tomographic ("CT") scan requested by the participants' doctor.

The purpose of this study is to collect information that will be used to determine if MSCs can be used to decrease inflammation and possibly slow down enlargement of the participants' aneurysm. The investigators will also be collecting blood samples to study special inflammatory cells that cause aneurysms as well as asking participants to have a "PET" (positron emission tomography) scan that can measure inflammation directly in the participants' aneurysm.

DETAILED DESCRIPTION:
This is a phase I, double blinded trial that will enroll 50 patients with Abdominal Aortic Aneurysms (AAA) measuring 3-5 cm in maximal transverse diameter (MTD). This study will assess the safety of MSCs in doses of 1 million MSCs/kg. or 3 million MSCs/kg. delivered intra-venously. This trial test the hypothesis that MSCs, in a dose dependent fashion, promote the frequency and immune suppressor function of CD4+CD25+ FoxP3+ T-regulatory cells and decrease AAA inflammation as measured by 18-fluorodeoxyglucose positron emission tomography/computed tomography (PET/CT). The primary safety endpoints will be incidence of treatment related adverse events accrued over 24 months. Efficacy measures are changes in frequency and immune suppressor function of Tregs, number and cytotoxic activity of CD4+/CD8+ CD28- T-cells, activated monocytes, and changes in aortic inflammation as measured by uptake of 18-FDG PET/CT compared to baseline. Incidence of surgical intervention, aneurysm related death, quality of life, and major adverse cardiac events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Be 40 and 85 years of age.
* Have diagnosis of noninflammatory degenerative infrarenal abdominal aortic aneurysms measuring 3-5 cm. in diameter by Computed Tomography (CT) scan.
* Females of childbearing potential must be willing to use one form of birth control for the duration of the study. Female participants must undergo a blood or urine pregnancy test at screening.

Exclusion Criteria:

* Inflammatory AAA defined by a thickened aortic wall and retroperitoneal fibrosis and adhesions of peritoneal organs, and elevated erythrocyte sedimentation rate or in the opinion of investigator.
* Mycotic AAA defined as saccular morphology, a positive blood culture, fever, or in the opinion of the investigator.
* Symptomatic, Saccular, or any AAA associated with thoracic aorta dilatation >5.0 cm.
* Infra-renal AAA associated with Marfan's or Ehlers-Danlos Syndrome or other connective tissue disorders.
* Common or external iliac artery aneurysm > 30 cm. in maximal transverse diameter.
* AAA due to dissection.
* Allergy to iodine contrast.
* History of cancer within the last 5 years, except basal cell skin carcinoma with clean border pathology report.
* Estimated glomerular filtration rate (eGFR) < 30mL/min.
* Any condition requiring immunosuppressant medications (e.g., for treatment of organ transplants, psoriasis, Crohn's disease, alopecia areata, rheumatoid arthritis, scleroderma, lupus).
* Acute coronary syndrome (ACS) in the last 30 days prior to enrollment.*
* Congestive heart failure (CHF) hospitalization within the last 30 days prior to enrollment.*
* HIV or Hepatitis C (HCV) positive.
* Contraindication to Computed Tomography or known allergy to contrast media.
* Any bleeding diathesis defined as an International Normalized Ratio (INR) 2.0 (off anticoagulation therapy) or history of platelet count less than 70,000 or hemophilia.
* Pregnant or breast-feeding women.
* Significant hepatic dysfunction (alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than 2 times normal).
* Life expectancy less than two years.
* Inability to provide written informed consent due to cognitive or language barriers (interpreter permitted).
* Presence of any clinical condition that in the opinion of the PI or the sponsor makes the patient not suitable to participate in the trial.

  * As defined by the standard definitions of CHF and ACS by the American Heart Association.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Murphy, MD BS, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Infusion of 1 Million Allogenic MSCs/kg: In a randomized fashion, the MSCs, in the appropriate dose, will be shipped to the performance site where the MSCs will be thawed, diluted and administered. The thawed MSCs with be administered within 4 hours to subjects in a monitored setting with telemetry and pulse oximetry. Patients will be premedicated with hydrocortisone and diphenhydramine. All subjects will be monitored throughout the infusion procedure with vital signs and pulse oximetry at 15 minutes prior to infusion and ending 2 hours post procedure. They will also be evaluated for clinical signs of pulmonary distress. All patients will be admitted overnight for continued observation. The patient will be examined the following day and discharged home.
  MSCs: Intravenous infusion of 1 million allogeneic MSCs/kg.
  MSCs: Intravenous infusion of 3 million allogeneic MSCs/kg
  Placebo: Intravenous infusion of Plasmalyte A (placebo)
- Intravenous Infusion of 3 Million Allogeneic MSCs/kg: In a randomized fashion, the MSCs, in the appropriate dose, will be shipped to the performance site where the MSCs will be thawed, diluted and administered.The thawed MSCs with be administered within 4 hours to subjects in a monitored setting with telemetry and pulse oximetry. Patients will be premedicated with hydrocortisone and diphenhydramine. All subjects will be monitored throughout the infusion procedure with vital signs and pulse oximetry at 15 minutes prior to infusion and ending 2 hours post procedure. They will also be evaluated for clinical signs of pulmonary distress. All patients will be admitted overnight for continued observation. The patient will be examined the following day and discharged home.
  MSCs: Intravenous infusion of 1 million allogeneic MSCs/kg.
  MSCs: Intravenous infusion of 3 million allogeneic MSCs/kg
  Placebo: Intravenous infusion of Plasmalyte A (placebo)
- Intravenous Infusion of Plasmalyte A (Placebo): In a randomized fashion, the Plasmalyte A will be shipped to the performance site where it will be thawed and administered. The Plasmalyte A will be administered within 4 hours to subjects in a monitored setting with telemetry and pulse oximetry as will be performed on active groups in order to protect the blinding of this study. Patients will be pre-medicated with hydrocortisone and diphenhydramine. All subjects will be monitored throughout the infusion procedure with vital signs and pulse oximetry at 15 minutes prior to infusion and ending 2 hours post procedure. They will also be evaluated for clinical signs of pulmonary distress. All patients will be admitted overnight for continued observation. The patient will be examined the following day and discharged home.
  MSCs: Intravenous infusion of 1 million allogeneic MSCs/kg.
  MSCs: Intravenous infusion of 3 million allogeneic MSCs/kg
  Placebo: Intravenous infusion of Plasmalyte A (placebo)
Period: Overall Study
Arm/Group | Intravenous Infusion of 1 Million Allogenic MSCs/kg | Intravenous Infusion of 3 Million Allogeneic MSCs/kg | Intravenous Infusion of Plasmalyte A (Placebo)
Started | 6 | 10 | 12
Completed | 0 | 0 | 0
Not Completed | 6 | 10 | 12
Not completed — Death | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Study terminated by VA DSMB due to low enrollment | 5 | 9 | 9
Not completed — Primary endpoint - endovascular aortic repair | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intravenous Infusion of 1 Million Allogenic MSC's/Kg: In a randomized fashion, the MSCs, in the appropriate dose, will be shipped to the performance site where the MSCs will be thawed, diluted and administered. The thawed MSCs with be administered within 4 hours to subjects in a monitored setting with telemetry and pulse oximetry. Patients will be premedicated with hydrocortisone and diphenhydramine. All subjects will be monitored throughout the infusion procedure with vital signs and pulse oximetry at 15 minutes prior to infusion and ending 2 hours post procedure. They will also be evaluated for clinical signs of pulmonary distress. All patients will be admitted overnight for continued observation. The patient will be examined the following day and discharged home.
  MSCs: Intravenous infusion of 1 million allogeneic MSCs/kg.
  MSCs: Intravenous infusion of 3 million allogeneic MSCs/kg
  Placebo: Intravenous infusion of Plasmalyte A (placebo)
- Total: Total of all reporting groups
Arm/Group | Intravenous Infusion of 1 Million Allogenic MSC's/Kg | Intravenous Infusion of 3 Million Allogeneic MSCs/kg | Intravenous Infusion of Plasmalyte A (Placebo) | Total
Number analyzed (Participants) | 6 | 10 | 12 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 3 | 9
  >=65 years | 2 | 8 | 9 | 19
Age, Continuous [Mean (Full Range); unit: years] | 64.17 [59 to 69] | 69 [65 to 75] | 67.75 [53 to 77] | 67.43 [53 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 10 | 12 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 10 | 12 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 6 | 10 | 11 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 10 | 12 | 28
AAA size 3.0 - 3.9 cm (max. transverse diameter) [Count of Participants; unit: Participants] | 2 | 7 | 5 | 14
AAA size 4.0 - 5.0 cm (max. transverse diameter) [Count of Participants; unit: Participants] | 4 | 3 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Changes in Circulating Inflammatory Cell Phenotypes as Measured by Mass Cytometry
Description: This trial will test the hypothesis that MSCs, in a dose dependent fashion (1 x 10^6 MSC/kg vs 3 x 10^6 MSC/kg) promote the frequency and immune suppressor function of Treg cells as measured by mass cytometry compared to baseline.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Intravenous Infusion of 1 Million Allogenic MSCs/kg | Intravenous Infusion of 3 Million Allogeneic MSCs/kg | Intravenous Infusion of Plasmalyte A (Placebo)
Number analyzed (Participants) | 6 | 10 | 12
cells | 21.2 (3.2) | 73.2 (6.9) | 0.1 (0.2)
Statistical Analysis 1: Comparison: Intravenous Infusion of 1 Million Allogenic MSCs/kg vs Intravenous Infusion of 3 Million Allogeneic MSCs/kg vs Intravenous Infusion of Plasmalyte A (Placebo); The primary statistical evaluation for Aim 1 will focus on the chronologically increasing counts of T-regulatory cells over time following MSC administration in both delivery groups. Using the pattern of increased counts with time and the standard deviation reported by Ito and colleagues in healthy subjects, 36 subjects provides 81.0% power to detect such a change.A p value of <0.05 will be considered significant; Test type: Superiority — These power estimates are based on linear regression of regulatory T-cell counts at each time point. These data will be summarized with the mean, median, standard deviation, standard error, minimum and maximum; p < 0.05, Regression, Cox — P value is adjusted for multiple comparisons; See above; Mean Difference (Final Values) = 81. — Estimates for the differences in the secondary endpoints will be used to perform a power estimation using a Monte Carlo simulation method

2. Secondary Outcome: Incidence of Treatment Related Adverse Events at 12 Months Post MSC Administration as Evidenced by the Investigator
Description: The safety of systemic administration of allogeneic MSCs will be measured by treatment-related adverse events over a period of 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Infusion of 1 Million Allogenic MSCs/kg | Intravenous Infusion of 3 Million Allogeneic MSCs/kg | Intravenous Infusion of Plasmalyte A (Placebo)
Number analyzed (Participants) | 6 | 10 | 12
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: All adverse events (treatment related or otherwise) were collected throughout each participants enrollment at Day 0 (study product infusion), Day 7, Day 12, Month 1, Month 6 and Month 12 time points.
Arm/Group | Intravenous Infusion of 1 Million Allogenic MSCs/kg | Intravenous Infusion of 3 Million Allogeneic MSCs/kg | Intravenous Infusion of Plasmalyte A (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/10 | 1/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/10 | 1/12
Other Adverse Events (participants affected / at risk) | 3/6 | 2/10 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Infusion of 1 Million Allogenic MSCs/kg (N=6) | Intravenous Infusion of 3 Million Allogeneic MSCs/kg (N=10) | Intravenous Infusion of Plasmalyte A (Placebo) (N=12)
Unanticipated Adverse Device Event (Product Issues) | 0 (0) | 0 (0) | 1 (1) — Study product sterility culture, pre-administration, was positive on Day 7. No adverse effects experienced by subject.
Prostatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis, acute, recurrent (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Critical Limb Threatening Ischemia (Vascular disorders) | 0 (0) | 2 (3) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (2)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation, new (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid volume overload (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1)
Congestive Heart Failure exacerbation (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1)
Anemia, recurrent (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pain, epigastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis externa, severe (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue, worsening (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Neck edema, significant (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Colitis with crypt micro-abscesses
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Infusion of 1 Million Allogenic MSCs/kg (N=6) | Intravenous Infusion of 3 Million Allogeneic MSCs/kg (N=10) | Intravenous Infusion of Plasmalyte A (Placebo) (N=12)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 1 (3) | 1 (1) | 0 (0)
Pancreatitis, acute, recurrent (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pain, abdominal (General disorders) | 3 (4) | 1 (1) | 1 (1)
Pain, back (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Pain, knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Lung nodule, new (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Colon Polyp Removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The major limitation of this trial is that it did not complete enrollment of the planned 36 subjects. This is because the trial was put on hold during the COVID pandemic and when the Richard Roudebush VAMV opened for elective procedures the VA Merit grant had expired.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT02846883/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT02846883/ICF_001.pdf